CLINICAL TRIAL: NCT03988530
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of the Safety, Efficacy and Pharmacokinetics of DPI-386 Nasal Gel for the Prevention and Treatment of Nausea Associated With Motion Sickness in Senior Subjects With Open-Label Follow-Up
Brief Title: Prevention and Treatment of Nausea Associated With Motion Sickness in Senior Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DPI-386-MS-24
Record Dates: First submitted 2019-06-06; First posted 2019-06-17 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Motion Sickness
Keywords: Anticholinergic; Scopolamine
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double-blinded placebo controlled for all treatment arms on Treatment Day 1. All DPI-386 Nasal Gel and placebo nasal gel vials are opaque and indistinguishable. The DPI-386 Nasal Gel and placebo nasal gels are identical in color and viscosity, and without identifiable smell. Treatment Days 2-4 are open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DPI-386 Nasal Gel (Active Comparator): DPI-386 Nasal Gel (0.2 mg / 0.12 g)
  Interventions: Drug: Scopolamine
- Placebo Nasal Gel (Placebo Comparator): placebo nasal gel (0.12 g)
  Interventions: Other: Placebo Nasal Gel

INTERVENTIONS:
Drug: Scopolamine — Subjects will self-administer DPI-386 Nasal Gel (0.2 mg / 0.12 g) or placebo nasal gel (0.12 g) on Treatment Day 1, and on Treatment Days 2 -4 all subjects will self administer DPI-386 Nasal Gel (0.2 mg / 0.12 g).
  Other Names: DPI-386 Nasal Gel
  Arms: DPI-386 Nasal Gel
Other: Placebo Nasal Gel — Placebo Nasal Gel (0.12g) twice a day on Treatment Day 1.
  Arms: Placebo Nasal Gel

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Safety, Efficacy and Pharmacokinetics of DPI 386 Nasal Gel for the Prevention and Treatment of Nausea Associated with Motion Sickness in Senior Subjects With Open-Label Follow-Up

DETAILED DESCRIPTION:
This Phase 3 clinical trial is a randomized, double-blind, placebo-controlled study with open-label follow-up to identify the safety, efficacy and pharmacokinetics of a repeated-dose regimen of DPI 386 nasal gel (intranasal scopolamine gel) for the prevention and treatment of nausea associated with motion sickness. The study will have two arms: DPI-386 nasal gel and placebo nasal gel for Treatment Day 1. Treatment Day 1 will include 50 subjects per arm, for a total of 100 subjects (n=100). All 100 subjects from Treatment Day 1 will receive open-label DPI-386 Nasal Gel for Treatment Days 2-4 (50 of these were originally randomized to receive placebo prior to receipt of the investigational product.).

Treatment Day 1 will be conducted aboard an ocean-going vessel to obtain data in an operationally relevant real world environment and within 30 days of Treatment Day 1, Treatment Days 2-4 will take place at the clinical site.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed and dated Informed Consent Form (ICF).
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 55 and over.
4. In good general health as evidenced by medical history with no recent history or current diagnosis of uncontrolled clinical problems as assessed by the Principal Investigator (PI) or qualified designee.
5. Ability to take intranasal medication and willingness to adhere to the study schedule and time constraints.
6. Agreement to adhere to the following lifestyle compliance considerations:

   * Refrain from consumption of grapefruit and any substance containing grapefruit for seven days prior to, during, and for seven days after the three Treatment Days.
   * Abstain from alcohol for 24 hours prior to first dose of study medication and during the three Treatment Days.

Exclusion Criteria:

1. Known allergic reactions to scopolamine or other anticholinergics.
2. Currently prescribed any of the following medication types and used within the specified washout periods below:

   * any form of scopolamine (including Transderm Scop®) (washout 5 days)
   * belladonna alkaloids (washout 2 weeks),
   * antihistamines (including meclizine) (washout 2 weeks),
   * tricyclic antidepressants (washout 2 weeks),
   * muscle relaxants (washout 4 days) and
   * nasal decongestants (washout 4 days)
3. Hospitalization or significant surgery requiring hospital admittance within the past six months.
4. Treatment with another investigational drug or other intervention within the past 30 days.
5. Having donated blood or plasma or suffered significant blood loss within the past 30 days.
6. Having any of the following medical conditions within the last two years or if any of the following medical conditions were experienced more than two years ago and are deemed clinically significant by the PI or qualified designee:

   * Significant gastrointestinal disorder, asthma, or seizure disorders.
   * History of cardiovascular disease.
   * History of vestibular disorders.
   * History of narrow-angle glaucoma.
   * History of urinary retention problems.
   * History of alcohol or drug abuse.
   * Nasal, nasal sinus, or nasal mucosa surgery.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
The efficacy endpoint is incidence of subjects who developed motion sickness and requested further treatment (i.e., subjects who received rescue medication). | During voyage on Treatment Day 1.
  The efficacy endpoint is incidence of subjects who developed motion sickness and requested further treatment (i.e., subjects who received rescue medication) during an 8 hour voyage on Treatment Day 1.
Safety of DPI-386 Nasal Gel compared to placebo nasal gel with an emphasis on cognitive adverse events. | During all four Treatment Days
  Safety endpoint is the incidence of adverse events.

SECONDARY OUTCOMES:
Severity of nausea as measured by the Visual Analog Scale (VAS) over the treatment period. | During Treatment Day 1 voyage.
  Respondents specify their degree of nausea by indicating a point along a continuous 100 mm line between two end-points; left one is for "No nausea" and the right one for "Very severe nausea". Scoring is based on the length from left point and a higher score means more severe degree of nausea (Spinks & Wasiak, 2011).
Safety in terms of cognition as measured by the Psychomotor Vigilance Task (PVT). | During Treatment Day 1 voyage
  The PVT is a neurocognitive assessment that measures alertness and tests sustained attention and reaction time. It was originally developed for sleep studies, and involves simple reaction time testing by requiring the participant to push a button as soon as the stimulus (a light) appears. After a response, the reaction time (in ms) is displayed. The inter-stimulus interval varies from two to 10 seconds, so it is not predictable, and the entire task takes 10 minutes (Dorrian, Rogers, & Dinges, 2005). There are also shorter versions which have been validated as reasonable substitutes for the 10 minute version, such as the five minute (Lamond, Dawson, & Roach, 2005)) and three minute versions (Grant, et al., (2017).
Describe the pharmacokinetics (PK) of a multi-dose schedule of DPI-386 Nasal Gel. | At time points -60, 30, 90, 120, 180, 330, 390, 450, 480 and 600 minutes during Treatment Days 2-4.
  PK parameters to be measured by Maximum Observed Plasma Concentration (Cmax)
Describe the pharmacokinetics (PK) of a multi-dose schedule of DPI-386 Nasal Gel. | At time points -60, 30, 90, 120, 180, 330, 390, 450, 480 and 600 minutes during Treatment Days 2-4.
  PK parameters to be measured by Time to Reach Maximum Observed Plasma Concentration (Tmax).
Describe the pharmacokinetics (PK) of a multi-dose schedule of DPI-386 Nasal Gel. | At time points -60, 30, 90, 120, 180, 330, 390, 450, 480 and 600 minutes during Treatment Days 2-4.
  PK parameters to be measured by Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: David R Helton, Study Director — Repurposed Therapeutics, Inc.
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
Publication